CLINICAL TRIAL: NCT05618093
Title: Use of Non-invasive Measurement of Cardiac Output and Stroke Volume to Assess Risk and Response to Treatment in Patients With PAH or CTEPH
Brief Title: Non-Invasive Measurement of Cardiac Output and Stroke Volume in PAH/CTEPH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study device no longer available
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-001981
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Arterial Hypertension; Chronic Thromboembolic Pulmonary Hypertension
Keywords: Pulmonary Arterial Hypertension; Chronic Thromboembolic Pulmonary Hypertension; PAH; CTEPH; Non-invasive Hemodynamics; Non-invasive Blood Pressure
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: This is a single center study to evaluate the use of non-invasive measurement of cardiac output and stroke volume to assess risk and response to treatment in patients with pulmonary arterial hypertension (PAH) and non- operable chronic thromboembolic pulmonary hypertension (CTEPH). We anticipate to enroll a total of 100 subjects at Ronald Reagan UCLA Medical Center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients diagnosed with PAH or CTEPH (Experimental): Patients with a confirmed diagnosis or suspected diagnosis of pulmonary arterial hypertension (PAH) or chronic thromboembolic pulmonary hypertension (CTEPH) prior to initiation or change in therapy.
  Interventions: Device: Non-invasive hemodynamic measurements

INTERVENTIONS:
Device: Non-invasive hemodynamic measurements — A patient profile will be set up in the Edwards EV1000 clinical platform by inputting the patient's demographic information. One or two Edwards ClearSight finger cuffs will be placed on the index, middle, and/or ring finger on one hand of the patient. A pressure controller will be secured by a forearm strap where the finger cuffs will be connected to the pressure controller. The pressure controller will be connected to the Edwards EV1000 clinical platform monitor. A heart reference sensor (HRS) will be connected to the pressure controller, a finger cuff, and to the patient at heart level. The Edwards EV1000 clinical platform will calibrate the finger probes, then record measurements for 10-30 seconds. If two finger probes are available, measurements will alternate between fingers.
  Other Names: Non-invasive blood pressure (NIBP)

SUMMARY:
Pulmonary arterial hypertension (PAH) and chronic thromboembolic pulmonary hypertension (CTEPH) are severe clinical conditions that, despite advances in therapeutics over the past 20 years, lead to serious morbidity and mortality. Guidelines on the diagnosis and treatment of pulmonary hypertension (PH) recommend the use of a multiparametric risk stratification tool to determine severity of disease, which should guide initial therapy and therapy modulation. This multiparametric risk stratification schema includes objective assessment of exercise capacity, right ventricular function and hemodynamic parameters in order to classify patients into severity categories. Cardiac index (CI) and right atrial pressure (RAP), measured via right heart catheterization (RHC), are the hemodynamic parameters used in risk assessment of PH. Arguably, stroke volume index (SVI) is the most important hemodynamic parameter for assessment of PH severity and there is currently no validated method for noninvasive measurement of cardiac output (CO), CI or SVI. Currently, a major obstacle in the field is that hemodynamic measurements are not obtained on a regular basis in the risk assessment and therapy modulation of patients with PAH and CTEPH. If a noninvasive method of hemodynamic measurement could be correlated with other objective measurements of risk assessment, it could become an invaluable tool in therapy initiation and modulation in the ambulatory setting.

This is a single center study to evaluate the use of non-invasive measurement of CO and stroke volume to assess risk and response to treatment in patients with PAH and non- operable CTEPH. We anticipate to enroll a total of 100 subjects at Ronald Reagan UCLA Medical Center.

A maximum of 10 hour in total for the study including the consent process, pre-procedure care, RHC procedure, and follow up visit. The initial visit will be approximately 4 hours with the RHC procedure itself will only be 20 minutes. Each follow up visit will be 1.5 hour.

Patients with known or suspected PAH or CTEPH will undergo a RHC as part of his or her standard of care. Three techniques of CO measurement will be performed sequentially at the time of the RHC.

The device that will be used is the Edwards ClearSight system and EV1000 clinical platform, a device that measures NIBP.

Patients will be followed over the period of 1 year every 3 months to obtain serial measurements for six-minute walk distance (6MWD), World Health Organization (WHO)/New York Heart Association Functional Class (FC), B-type natriuretic peptide (BNP) or N-terminal-pro hormone BNP (NT-proBNP), and non-invasive hemodynamic measurements. Additional visits will be scheduled to obtain the serial measurements one month prior and one month following if a patient is initiating or changing PH-specific therapy.

As this is a study looking at the feasibility of non-invasive measurement of cardiac output and stroke volume for risk assessment and response to therapy in pulmonary arterial hypertension (PAH) or chronic thromboembolic pulmonary hypertension (CTEPH), study personnel performing the study procedures will not be blinded to the clinical diagnosis and the management of the subject.

DETAILED DESCRIPTION:
This is a single center study to evaluate the use of non-invasive measurement of cardiac output and stroke volume to assess risk and response to treatment in patients with pulmonary arterial hypertension (PAH) and non- operable chronic thromboembolic pulmonary hypertension (CTEPH). We anticipate to enroll a total of 100 subjects at Ronald Reagan UCLA Medical Center.

After informed consent is obtained, the following procedure will be performed:

Patients with known or suspected pulmonary arterial hypertension (PAH) or chronic thromboembolic pulmonary hypertension (CTEPH) will undergo a right heart catheterization (RHC) as part of his or her standard of care. Three techniques of cardiac output (CO) measurement will be performed sequentially at the time of the RHC. The order of cardiac output testing will be randomized after informed consent is obtained and prior to the procedure. The operator performing the RHC procedure will be blinded to both the non-invasive blood pressure (NIBP) measurement and direct Fick cardiac output (CO) measurements while performing thermodilution cardiac output (CO) measurement.

The device that will be used is the Edwards ClearSight system and EV1000 clinical platform, a device that measures non-invasive blood pressure (NIBP).

Patients will be followed over the period of 1 year, up to every 3 months, to obtain serial measurements of six-minute walk distance (6MWD), World Health Organization (WHO)/New York Heart Association Functional Class (FC), and B-type natriuretic peptide (BNP) or N-terminal-pro hormone BNP (NT-proBNP) as part of standard of care. These serial measurements will be collected from the patient's medical record. Non-invasive hemodynamic measurements will be performed for research purposes. Additional visits will be scheduled to obtain the serial measurements one month prior and one month following if a patient is initiating or changing PH-specific therapy.

As this is a study looking at the feasibility of non-invasive measurement of cardiac output and stroke volume for risk assessment and response to therapy in pulmonary arterial hypertension (PAH) or chronic thromboembolic pulmonary hypertension (CTEPH), study personnel performing the study procedures will not be blinded to the clinical diagnosis and the management of the subject.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age.
* The patient must understand and sign informed consent form (ICF).
* Patients with a confirmed diagnosis or suspected diagnosis of pulmonary arterial hypertension (PAH) or chronic thromboembolic pulmonary hypertension (CTEPH) prior to initiation or change in therapy.
* PAH or CTEPH patients undergoing right heart catheterization (RHC) as part of their standard of care.

Exclusion Criteria:

* BMI < 20 or BMI > 35.
* Height less than 120 cm.
* Diagnosis of atrial fibrillation, aortic or mitral valve insufficiency or stenosis, or end-stage renal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
stroke volume (SV) | 12 months
  Stroke Volume (SV) is the volume of blood in millilitres ejected from the each ventricle due to the contraction of the heart muscle which compresses these ventricles.
stroke volume index (SVI) | 12 months
  Stroke Volume Index (SVI) relates SV to body surface area (BSA), thus relating heart performance to the size of the individual. The unit of measurement is millilitres per square metre (ml/m2).
cardiac output (CO) | 12 months
  Cardiac Output (CO) is the amount of blood the heart pumps from each ventricle per minute. It is usually expressed in litres per minute (L/min).
cardiac index (CI) | 12 months
  Cardiac index (CI) is the cardiac output proportional to the body surface area (BSA). The unit of measurement is litres per minute per square metre (L/min/m2).
systemic vascular resistance (SVR) | 12 months
  Systemic vascular resistance (SVR) refers to the resistance to blood flow offered by all of the systemic vasculature, excluding the pulmonary vasculature.
  The units for SVR are most commonly expressed as pressure (mmHg) divided by cardiac output (mL/min), or mmHg⋅min⋅mL^-1
blood pressure (BP) | 12 months
  The pressure of the blood in the circulatory system, often measured for diagnosis since it is closely related to the force and rate of the heartbeat and the diameter and elasticity of the arterial walls.
  Systolic Blood Pressure in mmHg Diastolic Blood Pressure in mmHg
heart rate (HR) | 12 months
  The number of heartbeats per unit of time, usually per minute.
  Measured in beats per minute (BPM)

SECONDARY OUTCOMES:
six-minute walk distance (6MWD) | 12 months
  The distance covered over a time of 6 minutes. This is used as the outcome by which to compare changes in performance capacity.
B-type natriuretic peptide (BNP) or N-terminal-pro hormone BNP (NT-proBNP) | 12 months
  B-type natriuretic peptide (BNP) is a hormone produced by your heart. N-terminal (NT)-pro hormone BNP (NT-proBNP) is a non-active prohormone that is released from the same molecule that produces BNP. Both BNP and NT-proBNP are released in response to changes in pressure inside the heart. These changes can be related to heart failure and other cardiac problems. Levels goes up when heart failure develops or gets worse, and levels goes down when heart failure is stable.
World Health Organization (WHO)/New York Heart Association Functional Class (FC) | 12 months
  The World Health Organization functional classification (WHO-FC) is a tool used to measure disease severity in patients with PAH whereby health care providers (HCPs) use patient reports of symptom experience and activity limitations to make their assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Jasuja, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Galie N, Channick RN, Frantz RP, Grunig E, Jing ZC, Moiseeva O, Preston IR, Pulido T, Safdar Z, Tamura Y, McLaughlin VV. Risk stratification and medical therapy of pulmonary arterial hypertension. Eur Respir J. 2019 Jan 24;53(1):1801889. doi: 10.1183/13993003.01889-2018. Print 2019 Jan. PMID 30545971
- [Result] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M; ESC Scientific Document Group. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Heart J. 2016 Jan 1;37(1):67-119. doi: 10.1093/eurheartj/ehv317. Epub 2015 Aug 29. No abstract available. PMID 26320113
- [Result] Raina A, Humbert M. Risk assessment in pulmonary arterial hypertension. Eur Respir Rev. 2016 Dec;25(142):390-398. doi: 10.1183/16000617.0077-2016. PMID 27903661
- [Result] Maron BA. Hemodynamics should be the primary approach to diagnosing, following, and managing pulmonary arterial hypertension. Can J Cardiol. 2015 Apr;31(4):515-20. doi: 10.1016/j.cjca.2014.09.021. Epub 2014 Sep 28. PMID 25742869
- [Result] D'Alonzo GE, Barst RJ, Ayres SM, Bergofsky EH, Brundage BH, Detre KM, Fishman AP, Goldring RM, Groves BM, Kernis JT, et al. Survival in patients with primary pulmonary hypertension. Results from a national prospective registry. Ann Intern Med. 1991 Sep 1;115(5):343-9. doi: 10.7326/0003-4819-115-5-343. PMID 1863023
- [Result] Sandoval J, Bauerle O, Palomar A, Gomez A, Martinez-Guerra ML, Beltran M, Guerrero ML. Survival in primary pulmonary hypertension. Validation of a prognostic equation. Circulation. 1994 Apr;89(4):1733-44. doi: 10.1161/01.cir.89.4.1733. PMID 8149539
- [Result] Weatherald J, Boucly A, Chemla D, Savale L, Peng M, Jevnikar M, Jais X, Taniguchi Y, O'Connell C, Parent F, Sattler C, Herve P, Simonneau G, Montani D, Humbert M, Adir Y, Sitbon O. Prognostic Value of Follow-Up Hemodynamic Variables After Initial Management in Pulmonary Arterial Hypertension. Circulation. 2018 Feb 13;137(7):693-704. doi: 10.1161/CIRCULATIONAHA.117.029254. Epub 2017 Oct 25. PMID 29070502
- [Result] Weatherald J, Boucly A, Launay D, Cottin V, Prevot G, Bourlier D, Dauphin C, Chaouat A, Savale L, Jais X, Jevnikar M, Traclet J, De Groote P, Simonneau G, Hachulla E, Mouthon L, Montani D, Humbert M, Sitbon O. Haemodynamics and serial risk assessment in systemic sclerosis associated pulmonary arterial hypertension. Eur Respir J. 2018 Oct 18;52(4):1800678. doi: 10.1183/13993003.00678-2018. Print 2018 Oct. PMID 30209196
- [Result] Yung GL, Fedullo PF, Kinninger K, Johnson W, Channick RN. Comparison of impedance cardiography to direct Fick and thermodilution cardiac output determination in pulmonary arterial hypertension. Congest Heart Fail. 2004 Mar-Apr;10(2 Suppl 2):7-10. doi: 10.1111/j.1527-5299.2004.03406.x. PMID 15073478
- [Result] Dupuis M, Noel-Savina E, Prevot G, Tetu L, Pillard F, Riviere D, Didier A. Determination of Cardiac Output in Pulmonary Hypertension Using Impedance Cardiography. Respiration. 2018;96(6):500-506. doi: 10.1159/000486423. Epub 2018 Feb 9. PMID 29428946
- [Result] Humbert M, Guignabert C, Bonnet S, Dorfmuller P, Klinger JR, Nicolls MR, Olschewski AJ, Pullamsetti SS, Schermuly RT, Stenmark KR, Rabinovitch M. Pathology and pathobiology of pulmonary hypertension: state of the art and research perspectives. Eur Respir J. 2019 Jan 24;53(1):1801887. doi: 10.1183/13993003.01887-2018. Print 2019 Jan. PMID 30545970
- [Result] Simonneau G, Montani D, Celermajer DS, Denton CP, Gatzoulis MA, Krowka M, Williams PG, Souza R. Haemodynamic definitions and updated clinical classification of pulmonary hypertension. Eur Respir J. 2019 Jan 24;53(1):1801913. doi: 10.1183/13993003.01913-2018. Print 2019 Jan. PMID 30545968
- [Result] Humbert M, Sitbon O, Yaici A, Montani D, O'Callaghan DS, Jais X, Parent F, Savale L, Natali D, Gunther S, Chaouat A, Chabot F, Cordier JF, Habib G, Gressin V, Jing ZC, Souza R, Simonneau G; French Pulmonary Arterial Hypertension Network. Survival in incident and prevalent cohorts of patients with pulmonary arterial hypertension. Eur Respir J. 2010 Sep;36(3):549-55. doi: 10.1183/09031936.00057010. Epub 2010 Jun 18. PMID 20562126
- [Result] Humbert M, Sitbon O, Chaouat A, Bertocchi M, Habib G, Gressin V, Yaici A, Weitzenblum E, Cordier JF, Chabot F, Dromer C, Pison C, Reynaud-Gaubert M, Haloun A, Laurent M, Hachulla E, Cottin V, Degano B, Jais X, Montani D, Souza R, Simonneau G. Survival in patients with idiopathic, familial, and anorexigen-associated pulmonary arterial hypertension in the modern management era. Circulation. 2010 Jul 13;122(2):156-63. doi: 10.1161/CIRCULATIONAHA.109.911818. Epub 2010 Jun 28. PMID 20585011
- [Result] Boucly A, Weatherald J, Savale L, Jais X, Cottin V, Prevot G, Picard F, de Groote P, Jevnikar M, Bergot E, Chaouat A, Chabanne C, Bourdin A, Parent F, Montani D, Simonneau G, Humbert M, Sitbon O. Risk assessment, prognosis and guideline implementation in pulmonary arterial hypertension. Eur Respir J. 2017 Aug 3;50(2):1700889. doi: 10.1183/13993003.00889-2017. Print 2017 Aug. PMID 28775050
- [Result] Benza RL, Gomberg-Maitland M, Miller DP, Frost A, Frantz RP, Foreman AJ, Badesch DB, McGoon MD. The REVEAL Registry risk score calculator in patients newly diagnosed with pulmonary arterial hypertension. Chest. 2012 Feb;141(2):354-362. doi: 10.1378/chest.11-0676. Epub 2011 Jun 16. PMID 21680644
- [Result] Benza RL, Miller DP, Gomberg-Maitland M, Frantz RP, Foreman AJ, Coffey CS, Frost A, Barst RJ, Badesch DB, Elliott CG, Liou TG, McGoon MD. Predicting survival in pulmonary arterial hypertension: insights from the Registry to Evaluate Early and Long-Term Pulmonary Arterial Hypertension Disease Management (REVEAL). Circulation. 2010 Jul 13;122(2):164-72. doi: 10.1161/CIRCULATIONAHA.109.898122. Epub 2010 Jun 28. PMID 20585012
- [Result] Benza RL, Miller DP, Barst RJ, Badesch DB, Frost AE, McGoon MD. An evaluation of long-term survival from time of diagnosis in pulmonary arterial hypertension from the REVEAL Registry. Chest. 2012 Aug;142(2):448-456. doi: 10.1378/chest.11-1460. PMID 22281797
- [Result] Benza RL, Miller DP, Foreman AJ, Frost AE, Badesch DB, Benton WW, McGoon MD. Prognostic implications of serial risk score assessments in patients with pulmonary arterial hypertension: a Registry to Evaluate Early and Long-Term Pulmonary Arterial Hypertension Disease Management (REVEAL) analysis. J Heart Lung Transplant. 2015 Mar;34(3):356-61. doi: 10.1016/j.healun.2014.09.016. Epub 2014 Sep 28. PMID 25447572
- [Result] Hoeper MM, Huscher D, Ghofrani HA, Delcroix M, Distler O, Schweiger C, Grunig E, Staehler G, Rosenkranz S, Halank M, Held M, Grohe C, Lange TJ, Behr J, Klose H, Wilkens H, Filusch A, Germann M, Ewert R, Seyfarth HJ, Olsson KM, Opitz CF, Gaine SP, Vizza CD, Vonk-Noordegraaf A, Kaemmerer H, Gibbs JS, Pittrow D. Elderly patients diagnosed with idiopathic pulmonary arterial hypertension: results from the COMPERA registry. Int J Cardiol. 2013 Sep 30;168(2):871-80. doi: 10.1016/j.ijcard.2012.10.026. Epub 2012 Nov 17. PMID 23164592
- [Result] Kylhammar D, Kjellstrom B, Hjalmarsson C, Jansson K, Nisell M, Soderberg S, Wikstrom G, Radegran G. A comprehensive risk stratification at early follow-up determines prognosis in pulmonary arterial hypertension. Eur Heart J. 2018 Dec 14;39(47):4175-4181. doi: 10.1093/eurheartj/ehx257. PMID 28575277
- [Result] Siedlecka J, Siedlecki P, Bortkiewicz A. Impedance cardiography - Old method, new opportunities. Part I. Clinical applications. Int J Occup Med Environ Health. 2015;28(1):27-33. doi: 10.13075/ijomeh.1896.00451. PMID 26159944
- [Result] De Maria AN, Raisinghani A. Comparative overview of cardiac output measurement methods: has impedance cardiography come of age? Congest Heart Fail. 2000 Mar-Apr;6(2):60-73. doi: 10.1111/j.1527-5299.2000.80139.x. PMID 12029189
- [Result] van Wolferen SA, Marcus JT, Boonstra A, Marques KM, Bronzwaer JG, Spreeuwenberg MD, Postmus PE, Vonk-Noordegraaf A. Prognostic value of right ventricular mass, volume, and function in idiopathic pulmonary arterial hypertension. Eur Heart J. 2007 May;28(10):1250-7. doi: 10.1093/eurheartj/ehl477. Epub 2007 Jan 22. PMID 17242010
- [Result] Galie N, Palazzini M, Manes A. Pulmonary arterial hypertension: from the kingdom of the near-dead to multiple clinical trial meta-analyses. Eur Heart J. 2010 Sep;31(17):2080-6. doi: 10.1093/eurheartj/ehq152. Epub 2010 May 26. No abstract available. PMID 20504865
- [Result] Humbert M, Sitbon O, Chaouat A, Bertocchi M, Habib G, Gressin V, Yaici A, Weitzenblum E, Cordier JF, Chabot F, Dromer C, Pison C, Reynaud-Gaubert M, Haloun A, Laurent M, Hachulla E, Simonneau G. Pulmonary arterial hypertension in France: results from a national registry. Am J Respir Crit Care Med. 2006 May 1;173(9):1023-30. doi: 10.1164/rccm.200510-1668OC. Epub 2006 Feb 2. PMID 16456139
- [Result] Peacock AJ, Murphy NF, McMurray JJ, Caballero L, Stewart S. An epidemiological study of pulmonary arterial hypertension. Eur Respir J. 2007 Jul;30(1):104-9. doi: 10.1183/09031936.00092306. Epub 2007 Mar 14. PMID 17360728